CLINICAL TRIAL: NCT00508339
Title: Functional Outcomes Following Limb Sparing Surgery for Soft Tissue Sarcoma and Pre-Operative Radiotherapy
Brief Title: Functional Outcomes Following Limb Sparing Surgery for Sarcoma Patients
Status: Withdrawn | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0111
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Sarcoma
Keywords: Soft Tissue Sarcoma; Limb Sparing Surgery; Toronto Extremity Salvage Score; Radiotherapy; Quality of Life; Questionnaire; Survey; TESS
MeSH Terms: conditions — Sarcoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with a diagnosis of soft tissue sarcoma.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Toronto Extremity Salvage Score (TESS) questionnaire.
  Other Names: Survey

SUMMARY:
Primary Objectives:

1. To classify the types of wound healing complications that occur after pre-operative radiation therapy and limb sparing resection for the treatment of soft tissue sarcomas of the extremity.
2. To evaluate the impact of each complication type on patient function and quality of life using the Toronto Extremity Salvage Score (TESS).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of soft tissue sarcoma with histopathologic confirmation.
2. Treatment protocol that includes pre-operative radiation therapy.
3. Treatment protocol that includes limb-sparing surgical resection.
4. Patient has received MD Anderson Cancer Center multidisciplinary care.
5. Patient must be at least three years post-operative.

Exclusion Criteria:

1. Previous radiotherapy to the local site.
2. Presence of regional or distant metastases.
3. Major medical co-morbidities (eg. cerebrovascular accident, congestive heart failure, concurrent malignancy) or disabilities unrelated to treatment for soft tissue sarcoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of soft tissue sarcoma.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Endpoints for this study will be anatomic site, histological subtype, primary wound closure, wound complication type, need for secondary operation and type of secondary operation. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Charles E. Butler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States